CLINICAL TRIAL: NCT01816438
Title: A French Non Interventional Multicentric Cohort Study in Patients With Colorectal Dysplasia in Intestinal Inflammatory Diseases
Brief Title: A French Non Interventional Multicentric Cohort Study in Patients With Colorectal Dysplasia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hôpital Edouard Herriot (Other)
Responsible Party: Principal Investigator, Jean Christophe Saurin, Professor, Hôpital Edouard Herriot
Other Study IDs: SFED N°100
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Hyperplasia; Dysplasia
Keywords: abnormal histological colorectal lesions
MeSH Terms: conditions — Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples Without DNA — pathological lesion slides
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- dysplasia or colorectal lesion: 300 patients

SUMMARY:
The main purpose is to describe clinical practices nowadays prospectively about patients with a dysplasia diagnosis or another histological lesions.

It will be identified colic situation during the initial colonoscopy after dysplasia diagnosis or atypical lesion.

Also the frequency and the type of monitoring conducted about these patients(surgical and endoscopic treatments).

The main criterion evaluation will be the surgical and endoscopic rates during the time.

The treatments offered such as surgical, endoscopic ones or none of them will be followed.

Finally, the outcome of these patients: stability, lesion disappearance, surgery or development of cancer with frequencies for each of them and relationships with histological abnormal colorectal lesion will be measured.

DETAILED DESCRIPTION:
A replay centralized pathological lesion slides corresponding to the different lesion will be done

ELIGIBILITY:
Inclusion Criteria:

* intestinal chronic inflammatory disease with at least one lesion such as hyperplasia or no dysplastic scalloped lesion, dysplastic scalloped lesion or low grade dysplasia or high grade dysplasia
* compliant patient
* endoscopic follow possible
* no settler cancer
* no serious pathology such as cancer

Exclusion Criteria:

* settler cancer
* serious pathology such as cancer
* no compliant patient
* endoscopic follow not possible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In France more than 40000 persons are concerned with a high risk of cancer because of ulcerative colitis for example
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-07; Primary Completion 2023-07 (Actual); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
endoscopies results | 4 years
  rates of surgery and endoscopic treatments frequency of development of a cancer or a high grade dysplasia according to a type of abnormal histological colorectal lesion

CONTACTS AND LOCATIONS:
Overall Officials: Saurin Jean Christophe, MSD, Principal Investigator — no affiliated
Locations (1):
- Edouard Herriot Hospital, Lyon, Auvergne-Rhône-Alpes, France